CLINICAL TRIAL: NCT01572324
Title: Phase II Study of Hepatic Arterial Infusion With Oxaliplatin and Fluorouracil in Patients With Unresectable Biliary Tract Carcinomas
Brief Title: Study of Hepatic Arterial Infusion to Treat Biliary Tract Carcinomas
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Peking University (Other)
Responsible Party: Principal Investigator, Xiaodong Wang, MD, MD, Peking University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PUCH12031308
Record Dates: First submitted 2012-04-04; First posted 2012-04-06 (Estimated); Last update posted 2017-01-04 (Estimated); Status verified 2017-01

CONDITIONS: Biliary Tract Cancer
Keywords: Cholangiocarcinoma; gallbladder cancer; Infusions; Intra-Arterial
MeSH Terms: conditions — Biliary Tract Neoplasms; Cholangiocarcinoma; Gallbladder Neoplasms | interventions — Oxaliplatin; Fluorouracil; Leucovorin; Capecitabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Arterial infusion (Experimental)
  Interventions: Drug: Oxaliplatin, Fluorouracil, Leucovorin, Capecitabine

INTERVENTIONS:
Drug: Oxaliplatin, Fluorouracil, Leucovorin, Capecitabine — HAI of Oxaliplatin and Fluorouracil: Oxaliplatin 130mg/m2 in split daily doses for 3 days, Fluorouracil 3000 mg/m2 in split daily doses for 3 days. Intraarterial Oxaliplatin plus intravenous Leucovorin 200 mg/m2 simultaneously over 2 hours followed by intraarterial Fluorouracil over 22 hours on Days 1-3 of each cycle, repeat every 21 days. After 4-6 cycles of HAI, maintenance treatment continue, Maintenance of Oral capecitabine 1,000 mg/m2 twice a day from days 1-14, Cycles were repeated every 21 days.
  Other Names: 1-OHP, Dacotin, Eloxatin, L-OHP;; 5-Fluorouracil,5FU;; Levofolinic acid,Folinic acid.

SUMMARY:
This Phase II clinical trial is to study the effectiveness and safety of continuous hepatic arterial infusion (HAI) of Oxaliplatin and Fluorouracil in Patients with Unresectable Biliary tract carcinomas, and to explore a better first-line treatment regimen for these patients.

ELIGIBILITY:
Inclusion Criteria:

* Patient must have histologically or cytologically confirmed Biliary tract carcinomas including intrahepatic, hilar cholangiocarcinoma and gallbladder cancer without evident liver metastasis.
* Patient must have locally advanced disease that is unresectable after review by the Hepatobiliary Surgery service
* Patient's Eastern Cooperative Oncology Group (ECOG) performance status must be =< 2 (Karnofsky >= 60%)
* Absolute neutrophil count >= 1,500/mcL
* Platelets >= 100,000/mcL
* Hemoglobin >= 90g/L
* Total bilirubin =< 2 X institutional upper limit of normal
* Aspartate aminotransferase (AST) (serum glutamic oxaloacetic transaminase [SGOT])/alanine aminotransferase (ALT) (serum glutamic pyruvate transaminase [SGPT]) =< 2.5 X institutional upper limit of normality
* Creatinine =< 1.5 X institutional upper limit of normal
* Albumin >= 30g/L
* Patient must be able to understand and willing to sign a written informed consent document

Exclusion Criteria:

* Patients who have had prior chemotherapy and other antitumor therapy treatment
* Patient who is receiving any other investigational agents
* Patient who have evident distant (M) disease;
* Patient who have a diagnosis of hepatic encephalopathy
* Patients who have a diagnosis of sclerosing cholangitis.
* Patients who have a diagnosis of Gilbert's disease.
* Patients who have clinical ascites
* Patient must not have any uncontrolled concurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, uncontrolled diabetes mellitus and hypertension, or psychiatric illness/social situations that would limit compliance with study requirements
* No other malignancy except localized basal cell or squamous cell skin cancer in the past 5 years
* Patient who is pregnant or lactating
* Patient Allergic to Iodine contrast medium
* Uncontrolled severe coagulation disorders (INR < 1.5 in patients not on warfarin therapy)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 37 (Actual)
Dates: Start 2012-03; Primary Completion 2015-10 (Actual); Study Completion 2016-04 (Actual)

PRIMARY OUTCOMES:
Response rates | 4 months
  Describe the overall response rate with a 95% confidence interval.

SECONDARY OUTCOMES:
Progress free survivial | 2 years
  Describe median PFS with a 95% confidence interval.
Toxicity of HAI | 1 months
  Toxicity as measured by NCI Common Toxicity Criteria
Overall survival | 3 years
  Describe median overall survival with a 95% confidence interval and estimate the overall survival rate at 12 and 24 months with 24 months with a 95% confidence interval.

CONTACTS AND LOCATIONS:
Overall Officials: Xiaodong Wang, MD, Principal Investigator — Peking University Cancer Hospital & Institute
Locations (1):
- Peking University Cancer Hospital, Beijing, Beijing Municipality, China